CLINICAL TRIAL: NCT00005798
Title: A Phase II Study of Cyclophosphamide, Thiotepa, and Carboplatin (CTC) as a Preparative Regimen for Autologous Hematopoietic Stem Cell Transplantation in Patients With Breast Cancer
Brief Title: Combination Chemotherapy Followed By Peripheral Stem Cell Transplantation in Treating Women With Breast Cancer
Acronym: CTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11072; IRB-3898 (Other: University of South Florida); NCI-G00-1760 (Other: NCI)
Record Dates: First submitted 2000-06-02; First posted 2004-04-02 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Carboplatin; Cyclophosphamide; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTC Conditioning Regimen (Other): Cyclophosphamide Thiotepa Carboplatin
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Thiotepa

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given at a dose of 267 mg/m2 in D5 W IV over one hour daily on days -6, -5, and -4. (Total dose 800 mg/m2)
  Other Names: Paraplatin(R)
Drug: Cyclophosphamide — Cyclophosphamide will be given at a dose of 2000 mg/m2 in NS IV over one hour daily on days -6, -5, and -4. (Total dose 6000 mg/m2)
Drug: Thiotepa — Thiotepa will be given at a dose of 167 mg/m2 in NS IV over one hour daily on days -6, -5, and -4. (Total dose 500 mg/m2 )

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation in treating women who have breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine long term remission rates as measured by disease free survival in women with breast cancer treated with cyclophosphamide, thiotepa, and carboplatin followed by autologous hematopoietic stem cell transplantation. II. Determine the safety and efficacy of this combination chemotherapy regimen in this patient population.

OUTLINE: Peripheral blood stem cells (PBSC) are collected. Patients sequentially receive cyclophosphamide IV over 1 hour, thiotepa IV over 1 hour, and carboplatin IV over 1 hour on days -6 to -4. PBSC are reinfused on day 0. Patients are followed at 3 months, 6 months, 1 year, and then annually thereafter.

PROJECTED ACCRUAL: At least 40 patients with 4-9 positive lymph nodes and at least 50 patients with 10 positive lymph nodes will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed breast cancer Stage II with greater than 3 positive axillary lymph nodes following standard induction chemotherapy, as well as surgery and/or radiation as clinically indicated Stage III following standard induction chemotherapy with an anthracycline based regimen, and surgery and/or radiation as clinically indicated Inflammatory carcinoma following standard induction chemotherapy with an anthracycline based regimen, and surgery and/or radiation as clinically indicated Stage IV metastatic disease that has demonstrated a complete response to an anthracycline containing regimen, or no evidence of disease after surgery or radiation Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 64 and under Sex: Female Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT/SGPT no greater than 2.5 times upper limit of normal No history of severe hepatic dysfunction Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No evidence of severe cardiac dysfunction Ejection fraction at least 50% by MUGA No major heart disease Essential hypertension controlled with medications allowed Pulmonary: DLCO at least 50% of normal No symptomatic obstructive or restrictive pulmonary disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No psychosocial disorder that would preclude study compliance No concurrent active infections No insulin dependent diabetes mellitus No uncompensated major thyroid or adrenal dysfunction No significant skin breakdown from tumor or other disease HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Prior total dose of doxorubicin or daunorubicin less than 450 mg/m2 unless endometrial biopsy shows less than grade 2 drug effect Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No concurrent nitroglycerin preparations for angina pectoris No concurrent antiarrhythmic drugs for major ventricular dysrrhythmias

Ages: 15 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 209 (Actual)
Dates: Start 1995-07; Primary Completion 2001-08 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
relapse-free survival | five years post transplant
  relapse free survival determined by the Kaplan-Meier product-limit method

SECONDARY OUTCOMES:
Rate of Grade III/IV toxicities | five years post transplant
  rate of grade III/IV toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Anasetti, MD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - Halifax Medical Center, Daytona Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida